CLINICAL TRIAL: NCT03577782
Title: Phase II Clinical Trial to Analyze the Safety and Efficacy of Vedolizumab Combined With Antiretroviral Therapy to Achieve Permanent Virological Remission in HIV-infected Subjects Without Previous Antiretroviral Therapy
Brief Title: Vedolizumab Treatment in HIV-Infected Subjects Without Previous Antiretroviral Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Luis F. Lopez-Cortes, Senior Researcher Andalusian Health System, Hospitales Universitarios Virgen del Rocío
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIS-VED-2017-01; 2018-000497-30 (EudraCT Number)
Record Dates: First submitted 2018-06-12; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: HIV Infections
Keywords: HIV; CD4+; T-cell; Reservoir; Cure; Antiretroviral therapy; Vedolizumab; Gut; Alpha4Beta7; gp120; Interruption
MeSH Terms: conditions — HIV Infections | interventions — vedolizumab

STUDY DESIGN:
Intervention Model Description: HIV-infected subjects with no previous ART will begin ART together with Vedolizumab infusions at week 0, 4, 8, 12, 16, 20 and 24 weeks. At this time point ART and Vedolizumab treatment will be interrupted. Patients will be followed up until week 48. ART will be resumed if CD4+ T-cell levels drop below 350 CD4+/μL and/or viral load increases above 10e5 HIV-RNA copies/mL (two consecutive measurements).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): HIV-infected subjects with no previous ART will begin ART together with Vedolizumab infusions at week 0, 4, 8, 12, 16, 20 and 24 weeks. At this time point ART and Vedolizumab treatment will be interrupted. Patients will be followed up until week 48. ART will be resumed if CD4+ T-cell levels drop below 350 CD4+/μL and/or viral load increase above 10e5 HIV-RNA copies/mL (two consecutive measurements).
  Interventions: Biological: Entyvio (Vedolizumab)

INTERVENTIONS:
Biological: Entyvio (Vedolizumab) — 1. Antiretroviral treatment consisting in Dolutegravir (Tivicay) (50mg) + Tenofovir alafenamide (TAF) (25mg) / Emtricitabina (FTC) (200mg) (Descovy), once daily during 24 weeks.
  2. Entyvio (Vedolizumab) (300mg), 7 intravenous infusions at week 0 (baseline) (concomitant with ART onset), 4, 8, 12, 16, 20 and 24.
  At week 24 ART and Vedolizumab administration will be interrupted. ART will be resumed if CD4+ T-cell levels drop below 350 CD4+/μL and/or viral load increase above 10e5 HIV-RNA copies/mL (two consecutive measurements).
  Patients will be followed up until week 48.

SUMMARY:
HIV cannot be eliminated and remains in the body despite the treatment that is used for HIV-infection called antiretroviral treatment (ART). Individuals undergoing ART interruption rapidly experience virus rebound in the blood. The current alternative therapeutic strategies to antiretroviral treatment have the aim to achieve the elimination of the virus in blood in the absence of ART. New drugs associated to ART that allow the elimination of the virus in the blood after ART withdrawn are needed. In monkeys infected with SIV, the analog of HIV, the virus has disappeared from the blood after administration of a compound and cessation of ART. There is an equivalent compound in humans called Vedolizumab. The aim of the present study is to research if Vedolizumab combined with ART, in subjects without previous ART, is able to eliminate the virus from the blood after ART is not taken.

DETAILED DESCRIPTION:
HIV cannot be eradicated and keep latent in anatomical and cellular reservoirs. In fact, patients undergoing antiretroviral treatment (ART) interruption rapidly experience plasma viral load rebound. The current alternative therapeutic strategies to antiretroviral treatment have the aim to achieve the eradication or permanent remission of plasma viral load, also known as functional cure, in the absence of ART, as occurs in persistent HIV controllers. In this scenario, new drugs associated to ART that allow the achievement of permanent plasma viral remission after ART withdrawn are needed.

The main targets of HIV infection are the memory CD4+ T-cells. This cell subset is mainly located in gut associated lymphoid tissue (GALT). These lymphocytes are recruited to the gut thanks to the expression of the integrin α4β7. The Env protein gp120 binds to α4β7 and enable the dissemination of HIV in the gut. At the same time the envelope of HIV is enriched in α4β7 coming from the plasma membrane of the host cells favoring its pathogenicity. Recently, the administration of a monoclonal antibody against α4β7 was shown to achieve significant protection for HIV transmission before and after low dose intravaginal inoculation of SIV in Rhesus Macaques. Surprisingly, long-term virological protection has been documented in SIV-infected macaques after ART interruption after administration and withdrawal of the monoclonal antibody against α4β7. The mechanisms through which this antibody has achieved the permanent remission of plasma viral load are not fully understood. The success of these findings in the simian model makes the antibody against α4β7 a good candidate as ART adjuvant with the aim to reach a functional cure and/or persistent virological remission in humans. Currently, there is a monoclonal antibody against α4β7 with known safety and security profiles in humans, this antibody is commercially available under the name of Vedolizumab. This antibody is used for the treatment of ulcerative colitis and Crohn Disease. In fact, there are already two clinical trials that are using Vedolizumab in HIV-infected patients (NCT02788175 y NCT03147859). In these clinical trials Vedolizumab is administered in the chronic phase of the infection in subjects with undetectable viral load during at least two years on ART. There are not clinical trials administering Vedolizumab in early stages of infection in naïve HIV-infected subjects for ART. Potentially, this strategy of early antibody treatment may increase the success of the therapy and decrease the time on ART of the individuals. The aim of the present clinical trial is to evaluate the safety and efficacy of Vedolizumab combined with ART to achieve permanent virological remission in naïve HIV-infected individuals after ART interruption.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with documented HIV-infection. Aged, 18 - 65 years.
* HIV-RNA >1x10e4 copies/mL.
* CD4+ T-cell counts >350 cells//μL
* To accept analytical ART interruption.

Exclusion Criteria:

* Presence of major resistance mutations to the antiretrovirals used.
* Active opportunistic infections.
* Pregnancy or breastfeeding
* Active hepatitis C or B virus infection.
* Active or latent tuberculosis not treated.
* Cirrhosis, portal hypertension and/or hypersplenism of any etiology.
* Current or past neoplasia susceptible to be treated with steroids, immunotherapy or chemotherapy.
* Abnormal laboratory measurements grade 3 or 4.
* Concomitant use of drugs with pharmacological interactions with the treatment of the study based on the technical data sheet of the products.
* Creatinine clearance <50mL/min.
* Any type of vaccination (e.g., hepatitis B virus, influenza…) two weeks before the beginning of the study.
* Cardiovascular disease (e.g., acute coronary syndrome, heart failure…).
* Neurological or neuro psychiatric disorder which symptoms may interfere with the safety and tolerability analysis.
* Alcohol abuse and/or drugs that may interfere with the study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women during pregnancy or breast-feeding will be excluded. Women must agree to use suitable contraception method (hormonal or barrier method of birth control; abstinence) before entry and during the study.
Enrollment: 12 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 48 weeks
  The number of adverse events and severity during Vedolizumab infusions and during all the follow up.
Plasma viral load rebound or remision after interrupting Vedolizumab infusions and ART | 48 weeks
  Quantitative plasma viral load (Roche HIV-1 RNA Viral Load Assay) measured before and after interrupting Vedolizumab infusions and ART.

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Ruiz-Mateos, PhD, Principal Investigator — Virgen del Rocio University Hospital
Locations (1):
- Virgen del Rocío University Hospital, Seville, Spain

REFERENCES:
- [Background] Pernas M, Tarancon-Diez L, Rodriguez-Gallego E, Gomez J, Prado JG, Casado C, Dominguez-Molina B, Olivares I, Coiras M, Leon A, Rodriguez C, Benito JM, Rallon N, Plana M, Martinez-Madrid O, Dapena M, Iribarren JA, Del Romero J, Garcia F, Alcami J, Munoz-Fernandez M, Vidal F, Leal M, Lopez-Galindez C, Ruiz-Mateos E. Factors Leading to the Loss of Natural Elite Control of HIV-1 Infection. J Virol. 2018 Feb 12;92(5):e01805-17. doi: 10.1128/JVI.01805-17. Print 2018 Mar 1. PMID 29212942
- [Background] Cicala C, Martinelli E, McNally JP, Goode DJ, Gopaul R, Hiatt J, Jelicic K, Kottilil S, Macleod K, O'Shea A, Patel N, Van Ryk D, Wei D, Pascuccio M, Yi L, McKinnon L, Izulla P, Kimani J, Kaul R, Fauci AS, Arthos J. The integrin alpha4beta7 forms a complex with cell-surface CD4 and defines a T-cell subset that is highly susceptible to infection by HIV-1. Proc Natl Acad Sci U S A. 2009 Dec 8;106(49):20877-82. doi: 10.1073/pnas.0911796106. Epub 2009 Nov 20. PMID 19933330
- [Background] Arthos J, Cicala C, Martinelli E, Macleod K, Van Ryk D, Wei D, Xiao Z, Veenstra TD, Conrad TP, Lempicki RA, McLaughlin S, Pascuccio M, Gopaul R, McNally J, Cruz CC, Censoplano N, Chung E, Reitano KN, Kottilil S, Goode DJ, Fauci AS. HIV-1 envelope protein binds to and signals through integrin alpha4beta7, the gut mucosal homing receptor for peripheral T cells. Nat Immunol. 2008 Mar;9(3):301-9. doi: 10.1038/ni1566. Epub 2008 Feb 10. PMID 18264102
- [Background] Guzzo C, Ichikawa D, Park C, Phillips D, Liu Q, Zhang P, Kwon A, Miao H, Lu J, Rehm C, Arthos J, Cicala C, Cohen MS, Fauci AS, Kehrl JH, Lusso P. Virion incorporation of integrin alpha4beta7 facilitates HIV-1 infection and intestinal homing. Sci Immunol. 2017 May 12;2(11):eaam7341. doi: 10.1126/sciimmunol.aam7341. PMID 28763793
- [Background] Byrareddy SN, Kallam B, Arthos J, Cicala C, Nawaz F, Hiatt J, Kersh EN, McNicholl JM, Hanson D, Reimann KA, Brameier M, Walter L, Rogers K, Mayne AE, Dunbar P, Villinger T, Little D, Parslow TG, Santangelo PJ, Villinger F, Fauci AS, Ansari AA. Targeting alpha4beta7 integrin reduces mucosal transmission of simian immunodeficiency virus and protects gut-associated lymphoid tissue from infection. Nat Med. 2014 Dec;20(12):1397-400. doi: 10.1038/nm.3715. Epub 2014 Nov 24. PMID 25419708
- [Background] Byrareddy SN, Arthos J, Cicala C, Villinger F, Ortiz KT, Little D, Sidell N, Kane MA, Yu J, Jones JW, Santangelo PJ, Zurla C, McKinnon LR, Arnold KB, Woody CE, Walter L, Roos C, Noll A, Van Ryk D, Jelicic K, Cimbro R, Gumber S, Reid MD, Adsay V, Amancha PK, Mayne AE, Parslow TG, Fauci AS, Ansari AA. Sustained virologic control in SIV+ macaques after antiretroviral and alpha4beta7 antibody therapy. Science. 2016 Oct 14;354(6309):197-202. doi: 10.1126/science.aag1276. PMID 27738167
- [Background] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, Van Assche G, Axler J, Kim HJ, Danese S, Fox I, Milch C, Sankoh S, Wyant T, Xu J, Parikh A; GEMINI 1 Study Group. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013 Aug 22;369(8):699-710. doi: 10.1056/NEJMoa1215734. PMID 23964932
- [Background] Sandborn WJ, Feagan BG, Rutgeerts P, Hanauer S, Colombel JF, Sands BE, Lukas M, Fedorak RN, Lee S, Bressler B, Fox I, Rosario M, Sankoh S, Xu J, Stephens K, Milch C, Parikh A; GEMINI 2 Study Group. Vedolizumab as induction and maintenance therapy for Crohn's disease. N Engl J Med. 2013 Aug 22;369(8):711-21. doi: 10.1056/NEJMoa1215739. PMID 23964933
- [Derived] Jimenez-Leon MR, Gasca-Capote C, Roca-Oporto C, Espinosa N, Sobrino S, Fontillon-Alberdi M, Gao C, Roseto I, Gladkov G, Rivas-Jeremias I, Neukam K, Sanchez-Hernandez JG, Rigo-Bonnin R, Cervera-Barajas AJ, Mesones R, Garcia F, Alvarez-Rios AI, Bachiller S, Vitalle J, Perez-Gomez A, Camacho-Sojo MI, Gallego I, Brander C, McGowan I, Mothe B, Viciana P, Yu X, Lichterfeld M, Lopez-Cortes LF, Ruiz-Mateos E. Vedolizumab and ART in recent HIV-1 infection unveil the role of alpha4beta7 in reservoir size. JCI Insight. 2024 Jul 9;9(16):e182312. doi: 10.1172/jci.insight.182312. PMID 38980725